CLINICAL TRIAL: NCT00742443
Title: A Double Blind, Within Patient, Placebo Controlled Trial to Assess the Efficacy of Juvista (Avotermin) in Conjunction With Scar Revision Surgery for the Improvement of Disfiguring Scars.
Brief Title: Juvista in Scar Revision Surgery of Disfiguring Scars
Acronym: Revise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Julia Cook (Clinical Trial Manager), Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RN1001-0091
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Cicatrix
Keywords: Scar Revision
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Active versus Placebo within patient
  Interventions: Drug: Juvista (avotermin)
- 2 (Other): Active vs. Placebo within patient
  Interventions: Drug: Juvista (avotermin)
- 3 (Other): Active vs. Active within patient
  Interventions: Drug: Juvista (avotermin)

INTERVENTIONS:
Drug: Juvista (avotermin) — 100ng/100µL Juvista administered to each linear centimetre of the margins of one wound segment by intradermal injection immediately after and then 24h after wound closure versus 100μL of placebo administered to each linear centimetre of the margins of the other wound segment by intradermal injection immediately after and then 24h after wound closure
  Other Names: RN1001, TGFβ3
  Arms: 1
Drug: Juvista (avotermin) — 250ng/100µL Juvista administered to each linear centimetre of the margins of one wound segment by intradermal injection immediately after and then 24h after wound closure versus 100μL of placebo administered to each linear centimetre of the margins of the other wound segment by intradermal injection immediately after and then 24h after wound closure
  Other Names: RN1001, TGFβ3
  Arms: 2
Drug: Juvista (avotermin) — 250ng/100µL Juvista administered to each linear centimetre of the margins of both wound segments by intradermal injection immediately after and then 24h after wound closure
  Other Names: RN1001, TGFβ3
  Arms: 3

SUMMARY:
This trial is to determine whether Juvista can prevent scar formation or improve the appearance of scars following scar revision surgery. The trial will involve comparing Juvista to placebo.

DETAILED DESCRIPTION:
Each year, over one hundred million people undergo elective or emergency surgery and are left with scarring. Of these, over half a million patients undergo scar revision surgery. These types of scars are usually disfiguring, aesthetically unpleasant and can cause complications such as severe itching, tenderness, pain, depression and disruption of daily activities which can lead to a diminished quality of life. There is a clinical need for treatments that reduce scarring, as current therapies are often ineffective or inadequate.

Results from previous clinical trials show that Juvista is effective in improving scars in young and elderly males and females. Juvista-treated wounds appear to heal with scars that are more similar to the surrounding skin, and are narrower and paler with a faster fading of redness compared to placebo and standard care alone. This study will confirm the effectiveness of Juvista (avotermin) in the improvement of scar appearance when applied to the wound margins of patients following scar revision surgery of disfiguring scars.

The study is a double blind, within patient, placebo controlled, randomised trial in male and female patients. Patients will be asked to attend 10 study visits and will be followed up post-surgery for 12 months.

The potential benefits to the patients taking part in the trial will be that their scar is revised by a plastic surgeon. This procedure should leave subjects with a less noticeable scar. The existing scar will be surgically removed and the resulting wound will be divided into two segments of equal length. In most patients, one segment will receive treatment with Juvista administered by intradermal injection, the other with placebo. A few patients will receive treatment with Juvista to both segments of the wound.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years who have provided written informed consent.
* BMI between 15 and 35 kg/m2
* Patients with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests specified in the trial protocol.
* If females of child bearing potential, patients must be using a highly effective method(s) of contraception and agree to do so from at least the screening visit until one month after administration of the final study dose.
* The scar area to be revised is disfiguring. To be considered disfiguring for this trial scars must have at least one of the following characteristics.
* Scar area 13 or more cm in length.
* Scar area at least 0.6 cm wide at widest part.
* Surface contour of scar area elevated or depressed on palpation.
* Scar area adherent to underlying tissue.
* Skin hypo-or hyper-pigmented in an area exceeding 39cm2.
* Skin texture abnormal (irregular, atrophic, shiny, scaly, etc.) in an area exceeding 39cm2.
* The scar to be revised is at least 12 months old.
* The investigator considers that the appearance of the scar area to be revised can be improved with surgery alone.
* The scar area is linear and suitable for revision by excision and direct closure.
* The scar area to be revised is symmetrical in appearance around the mid-line.
* The scar area to be revised is between 7 and 20cm in length.
* The scar area to be revised runs along a flat surface which is in the same focal plane and suitable for accurate medical photography.
* The scar is approved for entry into the trial by the Independent Expert Screening Panel.

Exclusion Criteria

* Patients who on direct questioning and / or physical examination, have evidence of any past or present clinically significant medical condition that would impair wound healing.
* Patients with a creatinine clearance (CLcr) of 80ml/min or less. Creatinine clearance will be determined from the serum creatinine level at pre-study screening using the following formula :
* CLcr = (140-age (years)) x weight(kg)/ 72 x serum creatinine (mg/dL) {x 0.85 for females}
* Patients with a skin disorder that is chronic or currently active.
* Patients who, in the opinion of the Investigator, have significant ongoing psychiatric disorders, which may interfere with the trial assessments / visits.
* Patients with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Patients who are taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Patients undergoing investigations or changes in management for an existing medical condition (excluding the scar for revision).
* Patients who are or who become pregnant up to and including Day 0 or who are lactating.
* In the opinion of the Investigator, a patient who is not likely to complete the trial.
* Patients who on direct questioning and physical examination have history or evidence of keloid scarring.
* Patients with scar areas for revision that cross a joint or are in close proximity to an anatomical structure, which could lead to distortion of the resultant scar or difficulty in taking photographs.
* Patients with additional scars less than 3cm away from the area to be revised.
* Patients with scars that require revision using Z-plasty, W-plasty or any other such techniques.
* Patients who are involved in ongoing litigation in connection with the scar to be revised.
* Patients who have had surgery in the area to be excised within one year of Day 0.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Global Scar Comparison Scale as assessed by an Independent Clinical Scar Assessment Panel using photographs of the treated scars. | 12 months post surgery

SECONDARY OUTCOMES:
Global Scar Comparison Scale assessed by the patient looking at their own scars. | 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: D A McGrouther, FRCS, MD, Principal Investigator — University of Manchester
Locations (47):
- BodyAesthetic Research Center, St Louis, Missouri, United States
- Denmark (3):
  - Grymer Privathospital, Aarhus
  - Odense Universitetshopital, Odense
  - Sollorod Privethospital, Primary Clinic, Hjortholmsvej 2C, Viruni
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Hôpital maternité de Metz, Metz
  - CHU Lapeyronie, Montpelliers
  - Hôpital Emile Muller, Service de chirurgie plastique, Mulhouse
- Germany (11):
  - Martin Luther Krankenhaus, Berlin
  - Unfallkrankenhaus Berlin, Zentrum für Schwerbrandverletzte mit Plastischer Chirurgie, Warener Strasse 7, Berlin
  - BG-Universitätsklinik Bergmannsheil GmbH, Bochum
  - St Josef und St Elisabeth Hospital, Klinik fur Dermatologie und Allergologie, Gundrunstrasse 56, Bochum
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Friedrich-Schiller-Universität Jena, Klinik für Dermatologie, Erfurter Strasse 35, Jena
  - Rotes-Kreuz-Krankenhaus Kassel, Kassel
  - BG - Unfallklinik Ludwigshafen, Ludwigshafen Am Main
  - Universitätsklinikum Schleswig-Holstein- Campus Lübec Plastische Chirurgie, Handchirurgie, Ratzeburger Allee 160, Lübeck
  - Klinikum Offenbach GmbH - Chirurgische Klinik III, Starkenburgring 66, Offenbach
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
- Hungary (6):
  - Fővárosi Önkormányzat Egyesített Szent István és Szent László Kórház-Rendelőintézet, Budapest
  - HM Állami Egészségügyi Központ, Budapest
  - Magyarországi Református Egyház Bethesda Gyermekkórháza Égéssérült Gyermekeket Ellátó Országos Központ, Budapest
  - Kenézy Kórház Rendelőintézet Egészségügyi Szolgáltató Kft., Debrecen
  - Miskolci Egészségügyi Központ, Miskolc
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Italy (5):
  - Università degli studi di Genova, Genova
  - Chirurgia Plastica e Ricostruttiva, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione S. Maugeri, U.O. DI CHIRURGIA PLASTICA E RICOSTRUTTIVA, Pavia
  - Chirurgia Plastica, Umberto I Policlinico di Roma, Rome
  - Ospedale di Circolo di Varese "Fondazione Macchi", Chirurgia Plastica, Varese
- Paula Stradina Clinical University Hospital, Riga, Latvia
- Poland (5):
  - 110 Szpital Wojskowy z Przychodnia, Elblag
  - Klinkia Chirurgii Plastycznej, Akademickie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Zespół Zakładów Opieki Zdrowotnej Zachodniopomorski, Gryfice
  - Wojewódzki Szpital Specjalistyczny im. Ludwika Rydygiera, os. Złotej Jesieni 1, Krakow
  - Wojskowy Instytut Medyczny Kliniczny Oddział Chirurgii Plastycznej,, Warsaw
- Spain (6):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Nuestra Señora del Perpetuo Socorro, Albacete
  - Hospital de la Santa Creu I Sant Pau, Departamento Cirugía Plástica, Barcelona
  - Hospital Clinic, Departament o Cirugia plástica, Barcelona
  - Ibermutuamur, Madrid
  - Hospital de Conxo-Complejo Hospitalario Universitario de Santiago de Compostela, Servicio de Cirugía plástica, Santiago de Compostela
- United Kingdom (5):
  - Queen Victoria Hospital (QVH) NHS Foundation Trust, East Grinstead, West Sussex
  - Selly Oak Hospital, Birmingham
  - Bristol Plastic Surgery, Bristol
  - Nuffield Health Bristol Hospital, Bristol
  - Renovo Clinical Trials Unit, 48 Grafton Street, Manchester